CLINICAL TRIAL: NCT04522674
Title: A Pilot Trial Evaluating the Feasibility of Using Platelet-Rich Plasma (PRP) for Treatment of Symptomatic Osteoarthritis of the Lumbar Facet Joint(s) of the Spine
Brief Title: Platelet-Rich Plasma (PRP) for Treatment of Symptomatic Lumbar Facet Syndrome of the Spine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-3066
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Platelet-Rich Plasma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous platelet rich plasma (Experimental): 0.5 mL of activated autologous PRP will be injected by fluoroscopic guidance into the affected lumbar facet joint (s) depending on the number of affected levels. A max of 4 joints will be injected per patient.
  Interventions: Biological: Autologous platelet rich plasma

INTERVENTIONS:
Biological: Autologous platelet rich plasma — 0.5 mL autologous platelet rich plasma into a symptomatic osteoarthritic lumbar facet to treat back pain caused by lumbar facet syndrome

SUMMARY:
The purpose of this study is to investigate the feasibility of standardized autologous platelet rich plasma injections into osteoarthritic lumbar facet joints to treat back pain and improve patient function.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of z-joint mediated low back pain
* Pain rating of ≥4/10 on a VAS scale
* Symptom duration of 3 or more months
* Failed conservative therapy (minimum of PT and pain medications)
* Have diagnosis of lumbar facet syndrome after MRI, X-ray, or CT imaging of any severity and a medial branch block with local anesthetic that confirms lumbar facet pathology.

Exclusion Criteria:

* Inability to undergo fluoroscopically guided procedures
* Current pregnancy
* Prior spinal surgery with hardware
* Intolerance to local anesthesia, contrast medium, or blood derivatives
* Local or systemic infection or spinal infection
* Irreversible coagulopathy
* Patients that require strict anticoagulation and cannot be off antiplatelet medication for at least a week
* Less than 18 years of age
* Corticosteroid shot within last 3 months into affected lumbar facet joint because of concern of damage to cartilage in the joint in that time period.
* Patients with workman compensation related back pain
* Patients with rheumatic cause of lumbar facet arthritis.
* Patients who have had a radiofrequency neurotomy of the nerves innervating their affected facet joints within the last year

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Change in pain Visual Analog Score with back flexion and at rest from baseline after intervention over time. | Baseline, immediately after intervention, 1 week, 1 month, and 3 months post intervention
  Pain as assessed from 0-10. Where 10 is severe pain and 0 is no pain. Improvement of pain by 50% after intervention is defined as treatment success
PROMIS Survey for Low Back Pain Function (PROMIS-29) | Baseline, immediately after intervention, 1 week, 1 month, and 3 months post intervention
  NIH validated PROMIS score for physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, pain interference, and pain intensity (PROMIS- 29 Profile v2.0). A higher PROMIS T-score represents more of the concept being measured.For negatively-worded concepts like Anxiety,a T-score of 60 is one SD worse than average.By comparison,an Anxiety T-score of 40 is one SD better than average.However,for positively-worded concepts like Physical Function-Mobility,a T-score of 60 is one SD better than average while a T-score of 40 is one SD worse than average.

SECONDARY OUTCOMES:
Length of enrollment of 10 patients and attrition rate | 3 months
  Determine percentage of patients who enroll in the study, how long it takes to enroll 10 patients, and attrition rate of patients in a 3 month time period
Safety as measured by number of subjects with at least one adverse event | 3 months
  Monitoring of adverse events such as bleeding, infection, allergy, neurologic deficits, and injection-related complications.
Degree of improvement in pain and function based on severity of lumbar facet OA. | 3 months
  Using the surveys from the primary outcome, the investigators plan to perform a subgroup analysis depending on the severity of lumbar facet OA as seen by imaging

CONTACTS AND LOCATIONS:
Overall Officials: Venu R Akuthota, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado School of Medicine Spine Center, Aurora, Colorado, United States